CLINICAL TRIAL: NCT00650091
Title: Prednisone, Azathioprine, and N-acetylcysteine: A Study That Evaluates Response in IPF
Brief Title: Evaluating the Effectiveness of Prednisone, Azathioprine, and N-acetylcysteine in Patients With IPF
Acronym: PANTHER-IPF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00020066; U10HL080413-03 (NIH)
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Prednisone; Azathioprine; NAC; N-acetylcysteine
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive N-acetylcysteine (NAC) for 60 weeks.
  Interventions: Drug: N-acetylcysteine (NAC)
- 2 (Placebo Comparator): Participants will receive placebo for 60 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — Participants will receive 600 mg of NAC three times a day.
  Arms: 1
Drug: Placebo — Participants will receive placebo each day.
  Arms: 2

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a long-term lung disease that affects an individual's ability to breathe. In this randomized, double-blind, placebo-controlled trial, we assigned patients with idiopathic pulmonary fibrosis who had mild-to-moderate lung-function impairment to one of three groups - receiving a combination of prednisone, azathioprine, and NAC (combination therapy), NAC alone, or placebo - in a 1:1:1 ratio.

DETAILED DESCRIPTION:
IPF is a disease with widespread and permanent scarring of lung tissue which eventually results in death. Individuals with IPF may experience breathing difficulties, cough, chest pain, and a decreased exercise capacity. Although the cause of IPF is unknown, it may be a result of an inflammatory response to an unknown substance. NAC, an antioxidant that is effective at loosening up mucus that forms in the lungs, may improve lung function. The purpose of this study is to evaluate the effectiveness of NAC at preventing the loss of lung function in people with IPF.

In the initial double-blind, placebo-controlled trial, subjects who have idiopathic pulmonary fibrosis with mild-to-moderate impairment in pulmonary function are randomly assigned to receive a three-drug regimen of prednisone, azathioprine, and acetylcysteine; acetylcysteine alone; or placebo.

After safety concerns were identified by the data and safety monitoring board, the three-drug regimen was stopped by the National Heart, Lung, and Blood Institute (NHLBI) on October 14, 2011, and a clinical alert was issued. After a brief period of interruption for modification of the protocol and approval by the institutional review boards, patients continued to be recruited for the acetylcysteine group and the placebo group and were followed for the pre-specified duration of 60 weeks.

Study visits will occur at baseline and Weeks 4, 15, 30, 45, and 60. At all study visits, a physical exam and blood collection will occur. At selected visits, the following study procedures will occur: lung function testing; urine collection; a 6-minute walk test, and questionnaires to assess health status, breathing, and quality of life. Participants will record medication usage and symptoms in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Forced vital capacity (FVC) greater than or equal to 50% of predicted value
* Diffusion capacity (DLCO) greater than or equal to 30% of predicted value
* Diagnosis of IPF by modified American Thoracic Society (ATS) criteria in the 48 months before study entry

Exclusion Criteria:

* History of clinically significant environmental exposure known to cause pulmonary fibrosis
* Diagnosis of connective tissue disease as the likely cause of the interstitial disease
* Extent of emphysema greater than the extent of fibrotic change (i.e., honeycombing, reticular changes) on high resolution computed tomography (HRCT) scan
* Forced expiratory volume in 1 second (FEV1)/FVC ratio less than 0.65 at the time of screening (post-bronchodilator)
* Partial pressure of arterial oxygen (PaO2) less than 55 mm Hg (less than 50 mm Hg at Denver study site)
* Residual volume greater than 120% predicted at the time of screening (post-bronchodilator)
* Evidence of active infection
* Significant bronchodilator response on screening spirometry, defined as change in FEV1 greater than or equal to 12% and absolute change greater than 200 mL OR change in FVC greater than or equal to 12% and absolute change greater than 200 mL
* Screening and baseline FVC measurements (in liters, post-bronchodilator) differing by 11%
* Listed for lung transplantation
* History of unstable or deteriorating cardiac disease
* Heart attack, coronary artery bypass, or angioplasty in the 6 months before study entry
* Unstable angina pectoris or congestive heart failure requiring hospitalization in the 6 months before study entry
* Uncontrolled arrhythmia
* Severe uncontrolled high blood pressure
* Known HIV or hepatitis C
* Known cirrhosis and chronic active hepatitis
* Active substance and/or alcohol abuse
* Pregnant or breastfeeding
* Women of childbearing potential who are not using a medically approved means of contraception
* Any clinically relevant lab abnormalities, including the following:

  1. Creatinine greater than twice the upper limit of normal (ULN)
  2. Hematology outside of specified limits

     1. White blood cells less than 3,500/mm3
     2. Hematocrit less than 25% or greater than 59%
     3. Platelets less than 100,000 mm3 at the time of screening
  3. Any of the following liver function test criteria above specified limits

     1. Total bilirubin greater than twice the ULN
     2. Aspartate (AST) or alanine aminotransferases (ALT) greater than 1.5 the ULN
     3. Alkaline phosphatase greater than three times the ULN
     4. Albumin less than 3.0 mg/dL at the time of screening
* Known hypersensitivity to study medication
* Any condition other than IPF that, in the opinion of the site PI, is likely to result in death in the 1 year after study entry
* Any condition that, in the judgment of the PI, might cause participation in this study to be detrimental or makes the person a poor candidate for the study

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin I Schwarz, MD, Study Chair — University of Colorado, Denver; Kevin Brown, MD, Principal Investigator — National Jewish Health; Rob Kaner, MD, Principal Investigator — Weill Medical College at Cornell University; Talmadge King, MD, Principal Investigator — University of California, San Francisco; Joe Lasky, MD, Principal Investigator — Tulane University; James Loyd, MD, Principal Investigator — Vanderbilt University; Fernando Martinez, MD, Principal Investigator — University of Michigan; Imre Noth, MD, Principal Investigator — University of Chicago; Ganesh Raghu, MD, Principal Investigator — University of Washington; Jesse Roman, MD, Principal Investigator — Emory University; Jay Ryu, MD, Principal Investigator — Mayo Clinic; John Belperio, MD, Principal Investigator — University of California, Los Angeles; Kevin Anstrom, PhD, Principal Investigator — Duke University; Gail Weinmann, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Jeffrey Chapman, MD, Principal Investigator — The Cleveland Clinic; Lake Morrison, MD, Principal Investigator — Duke University; Michael Kallay, MD, Principal Investigator — Highland Hospital; Steven Sahn, MD, Principal Investigator — Medical University of South Carolina; Marilyn Glassberg, MD, Principal Investigator — University of Miami; Milton Rossman, MD, Principal Investigator — University of Pennsylvania; John Fitzgerald, MD, Principal Investigator — University of Texas; Mary Beth Scholand, MD, Principal Investigator — University of Utah; Neil Ettinger, MD, Principal Investigator — St. Luke's Hospital; Danielle Antin-Ozerkis, MD, Principal Investigator — Yale University; Joao deAndrade, MD, Principal Investigator — University of Alabama at Birmingham; Ivan Rosas, MD, Principal Investigator — Brigham and Women's; Joseph Zibrak, MD, Principal Investigator — Beth Isreal-Deaconess; Gerald Criner, MD, Principal Investigator — Temple University; Maria Padilla, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (26):
- United States (26):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Highland Hospital - University of Rochester Medical Center, Rochester, New York
  - Duke Universtiy, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health Research Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Andrade J, Schwarz M, Collard HR, Gentry-Bumpass T, Colby T, Lynch D, Kaner RJ; IPFnet Investigators. The Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet): diagnostic and adjudication processes. Chest. 2015 Oct;148(4):1034-1042. doi: 10.1378/chest.14-2889. PMID 26111071
- [Derived] Durheim MT, Collard HR, Roberts RS, Brown KK, Flaherty KR, King TE Jr, Palmer SM, Raghu G, Snyder LD, Anstrom KJ, Martinez FJ; IPFnet investigators. Association of hospital admission and forced vital capacity endpoints with survival in patients with idiopathic pulmonary fibrosis: analysis of a pooled cohort from three clinical trials. Lancet Respir Med. 2015 May;3(5):388-96. doi: 10.1016/S2213-2600(15)00093-4. Epub 2015 Apr 15. PMID 25890798
- [Derived] Idiopathic Pulmonary Fibrosis Clinical Research Network; Martinez FJ, de Andrade JA, Anstrom KJ, King TE Jr, Raghu G. Randomized trial of acetylcysteine in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2093-101. doi: 10.1056/NEJMoa1401739. Epub 2014 May 18. PMID 24836309
- [Derived] Idiopathic Pulmonary Fibrosis Clinical Research Network; Raghu G, Anstrom KJ, King TE Jr, Lasky JA, Martinez FJ. Prednisone, azathioprine, and N-acetylcysteine for pulmonary fibrosis. N Engl J Med. 2012 May 24;366(21):1968-77. doi: 10.1056/NEJMoa1113354. Epub 2012 May 20. PMID 22607134
- See also: Click here for the Idiopathic Pulmonary Fibrosis Clinical Research Network web site. — http://www.ipfnet.org
- See also: Clinical Alert: Commonly used three-drug regimen for idiopathic pulmonary fibrosis found harmful — http://www.nlm.nih.gov/databases/alerts/2011_nhlbi_ifp.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial Study Design: Subjects are randomly assigned to receive a three-drug regimen of prednisone, azathioprine, and acetylcysteine; acetylcysteine alone; or placebo.
  Amended Study Design: The three-drug regimen was removed from the protocol due to safety concerns on 10/14/2011. Subjects are randomly assigned to acetylcysteine or placebo.
Pre-assignment Details: Participants in the Pred/AZA/NAC group were discontinued and not re-randomized in the amended study.
Groups:
- N-Acetylcysteine: Participants will receive N-acetylcysteine (NAC) for 60 weeks.
  N-acetylcysteine (NAC): Participants will receive 600 mg of NAC three times a day.
- Placebo: Participants will receive placebo for 60 weeks.
  Placebo: Participants will receive placebo each day.
- Pred/AZA/NAC: The prednisone dose was started at 0.5 mg per kilo- gram of ideal body weight and was tapered to 0.15 mg per kilogram during a period of 25 weeks.
  The azathioprine dose (maximum, 150 mg per day) was based on the patient's ideal weight, concurrent use of allopurinol, and thiopurine methyl-transferase (TPMT) activity. NAC was prescribed at 600 mg orally three times a day.
Period: Initial Study Design - Interim Analysis
Arm/Group | N-Acetylcysteine | Placebo | Pred/AZA/NAC
Started | 81 | 78 | 77
Completed | 81 | 78 | 77
Not Completed | 0 | 0 | 0
Period: Amended Study Design
Arm/Group | N-Acetylcysteine | Placebo | Pred/AZA/NAC
Started | 133 | 131 | 0 (Study Drug was discontinued for all subjects due to safety concerns.)
Completed | 110 | 111 | 0
Not Completed | 23 | 20 | 0
Not completed — Withdrawal by Subject | 12 | 11 | 0
Not completed — Physician Decision | 5 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Lung transplantation | 4 | 2 | 0
Not completed — Other | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 133 | 131 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (6.4) | 67.2 (8.2) | 67.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 59
  Male | 107 | 98 | 205

OUTCOME MEASURES:

1. Primary Outcome: Overall Change in Forced Vital Capacity
Description: Change from Baseline in Forced Vital Capacity at 60 weeks (units in liters)
Time Frame: Measured as the estimated change from baseline to Week 60
Population: Analysis population includes participants from the amended study design only.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
liters | -0.18 [-0.23 to -0.12] | -0.19 [-0.24 to -0.14]

2. Secondary Outcome: Disease Progression
Description: The time-to-death or a 10% decline in FVC will be defined as the time-to-disease progression.
  The 10% decline in FVC from enrollment must be confirmed on 2 consecutive visits no less than 6 weeks apart. For subjects with 2 consecutive visits with a 10% decline in FVC, the time-to-disease progression will be defined as the time interval between enrollment and the initial visit with a 10% FVC decline.
Time Frame: Measured at Week 60
Population: Analysis population includes participants from the amended study design only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
percentage of participants | 27.1 [20.1 to 36.0] | 26.5 [19.5 to 35.4]

3. Secondary Outcome: Acute Exacerbations
Description: The following 3 criteria will define acute exacerbations in subjects with acute worsening of their respiratory conditions:
  1. Clinical (all of the following required): A) Unexplained worsening of dyspnea or cough within 30 days, triggering unscheduled medical care (e.g., emergency room, clinic, study visit, hospitalization). B) No clinical suspicion or overt evidence of cardiac event, pulmonary embolism, or deep venous thrombosis to explain acute worsening of dyspnea. C) No pneumothorax.
Time Frame: Measured at Week 60
Population: Analysis population includes participants from the amended study design only.
Measure: Number; unit: events
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
events | 3 | 3

4. Secondary Outcome: Respiratory Infections
Time Frame: Measured at Week 60
Population: Analysis population includes participants from the amended study design only.
Measure: Number; unit: events
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
events | 6 | 6

5. Secondary Outcome: Number of Participants With Maintained Forced Vital Capacity Response
Description: Maintained forced vital capacity response was a binary variable taking on a value of 1 for participants with higher FVC % predicted at week 60 compared to baseline.
Time Frame: Measured at Week 60
Population: Analysis population includes participants from the amended study design only.
Measure: Number; unit: participants
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
participants | 29 | 35

6. Post Hoc Outcome: Change in Forced Vital Capacity
Description: Change from Baseline in Forced Vital Capacity at 15, 30, 45, and 60 weeks (units in liters)
Time Frame: Baseline, 15, 30, 45, 60 week
Population: Analysis population includes participants from the amended study design only.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 133 | 131
liters
  15 week | -0.07 (0.19) | -0.04 (0.19)
  30 week | -0.07 (0.20) | -0.08 (0.25)
  45 week | -0.15 (0.25) | -0.15 (0.30)
  60 week | -0.16 (0.26) | -0.15 (0.30)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for amended study only.
Groups:
- Initial Study: Pred/AZA/NAC: Participants will receive prednisone, azathioprine, and N-acetylcysteine (NAC) for 60 weeks.
- Initial Study: Placebo: Placebo: Participants will receive placebo each day.
Arm/Group | N-Acetylcysteine | Placebo | Initial Study: Pred/AZA/NAC | Initial Study: Placebo
Serious Adverse Events (participants affected / at risk) | 25/133 | 20/131 | 24/77 | 8/78
Other Adverse Events (participants affected / at risk) | 123/133 | 117/131 | 68/77 | 61/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=133) | Placebo (N=131) | Initial Study: Pred/AZA/NAC (N=77) | Initial Study: Placebo (N=78)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (6) | 8 (9) | 2 (3)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5) | 4 (4) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intersticial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Fever (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=133) | Placebo (N=131) | Initial Study: Pred/AZA/NAC (N=77) | Initial Study: Placebo (N=78)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (44) | 32 (39) | 13 (15) | 18 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 26 (29) | 11 (12) | 10 (11)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 8 (10) | 9 (12) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 27 (31) | 26 (31) | 10 (11) | 10 (11)
Bronchitis (Infections and infestations) | 15 (26) | 13 (15) | 6 (6) | 6 (8)
Sinusitis (Infections and infestations) | 17 (22) | 10 (12) | 4 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 10 (13) | 11 (15) | 4 (6) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 18 (19) | 15 (18) | 6 (7) | 7 (8)
Nausea (Gastrointestinal disorders) | 14 (14) | 7 (9) | 10 (14) | 4 (4)
Constipation (Gastrointestinal disorders) | 12 (13) | 4 (4) | 2 (2) | 4 (4)
Fatigue (General disorders) | 9 (9) | 9 (9) | 8 (9) | 6 (6)
Oedema peripheral (General disorders) | 9 (11) | 6 (6) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (13) | 2 (2) | 5 (8)
Headache (Nervous system disorders) | 12 (14) | 12 (12) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 8 (9) | 8 (10) | 5 (7) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No